CLINICAL TRIAL: NCT06322225
Title: Construction and Demonstration of Accurate Prevention and Treatment System for Colorectal Tubular Adenoma
Brief Title: Establishment of Big Data Platform and Biobank for Colorectal Tubular Adenoma Lesions
Status: Not yet recruiting | Type: Observational
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Collaborators: National Key Research and Development Program of China (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2023YFC2507401
Record Dates: First submitted 2024-03-06; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Colorectal Tubular Adenoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral venous blood, urine, stool and adenoma tissue will be collected
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Colorectal tubular adenoma is the most common precancerous lesion of colorectal cancer, and the point is that its precise prevention and treatment can reduce the incidence of colorectal cancer.However, the epidemiological characteristics of colorectal tubular adenoma in China are unclear, the rate of missed diagnosis by colonoscopy is high, and the existing diagnosis and treatment techniques are lack of unified quality control standards,which makes it difficult to diagnose and achieve accurate prevention and control. How to improve the precise prevention and treatment of colorectal tubular adenoma and reduce the incidence of colorectal cancer is a major clinical scientific problem that needs to be solved urgently. For this purpose, this study was conducted in colorectal guided by the needs of accurate prevention and treatment of tubular adenoma lesions,and a multi-center colorectal tubular adenoma data management platform and a high-risk population database covering a full range of data including demographic characteristics, lifestyle factors, clinical information, endoscopic data and pathological images were established, biological sample databases of patients with pathological changes and high-risk populations were established, and data quality control and sample quality control standards were formulated standards-based.

The pathological prediction model and accurate risk assessment system of colorectal tubular adenoma were constructed by the pathological database.

ELIGIBILITY:
Inclusion Criteria:

Voluntarily sign informed consent; Colorectal tubular adenoma was diagnosed according to JSGE clinical guidelines They are between 18 and 70 years old

Exclusion Criteria:

Refuse to sign the informed consent Patients who were judged by the investigator to be unsuitable for participation in this study.

The diagnosis is not tubular adenoma of colorectal or other adenomas according to JSGE clinical guidelines Age < 18 or > 70

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: There were 30,000 patients diagnosed with colorectal tubular adenoma in our hospital and several research centers
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical information such as demographic characteristics, clinical data, endoscopy and pathological images | 2024.05-2026.12
  Through the collection of clinical data and biological samples, we established a tubular adenoma big data platform and biobank, and established a precision prevention and treatment system for tubular adenoma

IPD SHARING:
Plan to Share IPD: Undecided